CLINICAL TRIAL: NCT04026269
Title: Clinical Efficacy of MOAP Regimen for Relapsed/Refractory Classical Hodgkin's Lymphoma as a Rescue Therapy After Ineffective Treatment of Additional Low-dose Decitabine to Anti-PD-1 Antibody Camrelizumab
Brief Title: Clinical Efficacy of MOAP Regimen for Relapsed/Refractory cHL as a Rescue Therapy After DP Regimen
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Han weidong (Other)
Responsible Party: Sponsor-Investigator, Han weidong, Principal Investigator, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-043
Record Dates: First submitted 2019-07-18; First posted 2019-07-19 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Hodgkin Lymphoma
Keywords: MOAP; Relapsed/Refractory; Hodgkin Lymphoma; DP;
MeSH Terms: conditions — Hodgkin Disease; Recurrence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MOAP treatment (Experimental): Chlormethine Hydrochloride Injection 10mg d1,8 iv Vindesine Sulfate for Injection 4mg d1,8 iv Doxorubicin Hydrochloride Injection 25mg/m2 d1,8 iv Prednisone Acetate Tablets 1-1.5mg/kg/d d1-10 po 28 days/Cycle
  Interventions: Drug: MOAP

INTERVENTIONS:
Drug: MOAP — the new chemotherapy regimen for r/r cHL

SUMMARY:
The DP regimen, low-dose decitabine combined with SHR-1210, is the new treatment for relapsed or refractory classical Hodgkin's Lymphoma. Though the CR rate of this regimen is impressively high, which is verified more than 70% in our I/II phase study, there are also lots of patients cannot benefit from this treatment. On top of that, as the increasing utilization of mono-therapy or combination treatment with the immune checkpoint blockade (ICB), the adverse reactions associated with immunotherapy make it unavailable in parts of patients. The application of MOAP regimen to patients, who have a progressive disease after DP regimen, can bring high CR rate. MOAP can be the a rescue treatment for cHL resisted to DP treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have histological confirmation of relapsed or refractory Hodgkin lymphoma (HL).
2. 13 to 70 years of age.
3. ECOG performance of less than 2.
4. Life expectancy of at least 3 months.
5. Subjects with lymphoma must have at least one measureable lesion >1 cm as defined by lymphoma response criteria.
6. Subjects must have received at least two prior chemotherapy regimen and four cycle of DP regimen, and must be off therapy for at least 4 weeks prior to Day 1. Subjects with autologous hematopoietic stem-cell transplantation are eligible which must be more than 3 months.
7. Subjects must have adequate marrow, live, renal and heart functions.

Exclusion Criteria:

1. Subjects with any autoimmune disease or history of syndrome that requires corticosteroids or immunosuppressive medications.
2. Serious uncontrolled medical disorders or active infections, pulmonary infection especially.
3. Active alimentary tract hemorrhage or history of alimentary tract hemorrhage in 1 month .
4. Prior organ allograft.
5. Women who are pregnant or breastfeeding.
6. Women with a positive pregnancy test on enrollment or prior to investigational product administration.
7. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness.

Ages: 13 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-07-30 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
CRR assess by investigators per the 2014 Lugano classification | 3 years
  Time measured from the day of first documented PR or CR to the date of first rate of subjects achieved complete response in all evaluable subjects
Number of Subjects with treatment-related adverse events (AEs) | 2 years
  Incidence, nature, and severity of adverse events graded according to the NCI CTCAE v4.03.
duration of CR | 5 years
  Time measured from the day of first documented CR to the date of first documented progression, or death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Biotherapeutic Department of Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Study Protocol